CLINICAL TRIAL: NCT03686761
Title: Periodontal Changes and Gingival Soft Tissue Healing Following Mid Maxillary Distraction in Cleft Lip and Palate Patients
Brief Title: Periodontal Changes Following Mid Maxillary Distraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Ibrahim Madi, Principle investigator, University of Alexandria
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00010556
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Cleft Lip and Palate; Periodontal Pocket; Attachment Loss, Periodontal
Keywords: Inflammation; Healing; Distraction; Periodontium
MeSH Terms: conditions — Cleft Lip; Periodontal Pocket; Periodontal Attachment Loss; Inflammation

STUDY DESIGN:
Intervention Model Description: Surgical distraction was performed in 20 cleft lip and palate (CLP) subjects with class III malocclusion, gingival GCF were collected from teeth neighboring the osteotomy site and from premolars of the opposite arch as control.
Masking Description: The clinical assessment was not masked , however, the histological and biomarker examination were send to blind investigator not directly involved in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental): A Involvement with the osteotomy site of the surgery, osteotomy was performed then GCF were collected from teeth neighboring the
  Interventions: Procedure: A Involvement with the osteotomy site of the surgery
- Control (Active Comparator): Involvement with the osteotomy site of the surgery, surgical osteotomy was performed then GCF were collected from teeth away from the osteotomy site
  Interventions: Procedure: A Involvement with the osteotomy site of the surgery

INTERVENTIONS:
Procedure: A Involvement with the osteotomy site of the surgery — A Involvement with the osteotomy site of the surgery

SUMMARY:
To evaluate the health status of the periodontium and dentition at the distraction osteogenesis site in CLP subjects using mid maxillary distraction (MMD).

DETAILED DESCRIPTION:
Segmental forward maxillary distraction osteogenesis(DO)was performed. Distractor connecting buccal molar segments to the anterior maxilla was kept for 7 days. Then distraction was performed till overcorrection and consolidated for 3-months. Periodontal clinical parameters were recorded at baseline, 3 and 6-months postoperatively. Gingival crevicular fluid was collected . Soft tissue healing was evaluated clinically and histologically after distraction.

ELIGIBILITY:
Inclusion Criteria:

* Severe maxillary hypoplasia and negative anterior overjet

Exclusion Criteria:

* Systemic disease

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Measurement of periodontal inflammatory mediators | 7 days
  periodontal inflammatory mediators IL-1β

SECONDARY OUTCOMES:
Measurement of periodontal inflammatory mediators TNF- α | 7 days
  periodontal inflammatory mediators TNF- α
Assessment of periodontal probing depth | 3 and 6 month
  probing depth measurement
Assessment of clinical attachment loss | 3 and 6 month
  clinical attachment loss measurement
Assessment of periodontal clinical parameters | 3 and 6 month
  Gingival index evaluation GI

OTHER OUTCOMES:
Evaluating the gingival histological changes | 2 and 4 weeks
  histological examination of the soft tissue

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Madi, Principal Investigator — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No